CLINICAL TRIAL: NCT00445029
Title: Pathophysiological Study of Allergic Contact Dermatitis to Para-Phenylenediamine (PPD). Analysis of Cellular and Molecular Targets in Skin Inflammation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Other Study IDs: 2006.435
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Allergic Contact Dermatitis
Keywords: Allergic contact dermatitis; para-phenylenediamine; effector cells; regulatory cells; pathophysiology
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The current knowledge of the pathophysiology of allergic contact dermatitis is based on the murine model. In this model, CD8+ T cells are effector cells, and CD4+ T cells regulate the response by limiting the expansion of CD8+ T cells. The goal of this study is to characterize the pathophysiology of contact dermatitis, with patients allergic to para-phenylenediamine (PPD).

We suppose that the CD8+ T cells are the effectors of the allergic contact dermatitis, although the regulator cells belong to the LT CD4+ population. We will test our hypothesis on blood samples, and cutaneous biopsies of patients allergic to PPD.

ELIGIBILITY:
Inclusion Criteria:

For both groups:

* Patients aged from 18 to 65 years old.
* Both genders eligible for study.
* Female participants must use a contraceptive method.
* Feasibility of patch testing.
* Participants must be able to understand and sign the Informed Consent, and comply with all aspects of the protocol.
* Patients must be registered in a social security system or with a health insurance coverage

   First group: allergic patients
* Patients with allergic contact dermatitis to para-phenylenediamine (PPD) based on a history of PPD contact dermatitis and positive PPD patch tests.

   Second group : healthy volunteers
* No history of PPD allergic contact dermatitis, with a negative PPD patch test.

Exclusion Criteria:

* Pregnant or lactating women.
* Evolutive skin disease on the testing zone (lower back).
* Patients with a clinically significant disease (chronic, recurrent or active).
* Systemic corticotherapy or immunosuppressive treatment during the previous month, or local corticoid treatment the week before the patch testing.
* Local or systemic drug use which interacts with the outcome measures.
* Exposure to sun or UV radiations, 15 days before the patch testing.
* Patients deprived of their civic rights, in custody, or subject to a tutorial, judiciary or administrative decision.
* Patients subject to a protection measure.
* Patients in a critical medical situation.
* Patients with a personal situation judged by the investigator as unlikely to be compatible with optimal participation in the study, or which could constitute a risk for the patient.
* Linguistic barrier or psychological profile preventing the patient from signing the consent form.
* Patient still in an exclusion period following the participation in another clinical trial.
* Patients having earned more than 4500€ in indemnities for participation in clinical trials during the previous 12 months, including this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Nicolas, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Jean-François Nicolas, Lyon, France